CLINICAL TRIAL: NCT02744560
Title: Effect of Spirulina on Liver Iron Concentration in Beta Thalassemic Children With Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Elshanshory, head of pediatric hematology and oncology unit, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3026/01/15
Record Dates: First submitted 2016-04-16; First posted 2016-04-20 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

ARMS (1):
- patients (Experimental): 30 multitransfused beta thalassemic children infected with hepatitis C virus diagnosed by serological detection of HCV-antibodies and HCV RNA by polymerase chain reaction will be given Spirulina in a dose of 250 mg/kg/day orally for 3 months.
  Interventions: Dietary Supplement: spirulina

INTERVENTIONS:
Dietary Supplement: spirulina — Spirulina in a dose of 250 mg/kg/day will be given orally for 3 months.

SUMMARY:
Thalassemics can develop liver fibrosis because of iron overload and hepatitis C infection. The latter is the main risk factor for liver fibrosis in transfusion dependent thalassemics. Excess liver iron is clearly recognized as a co factor for the development of advanced fibrosis in patients with hepatitis virus C infection. Magnetic resonance imaging represents the most available noninvasive technique to assess the level of iron in the liver.there is evidence that suggests Spirulina may help to protect against liver damage, cirrhosis and liver failure in those with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* multitransfused beta thalassemic children with super added hepatitis C virus (HCV) infection diagnosed by serological detection of HCV antibodies and HCV RNA by polymerase chain reaction.

Exclusion Criteria:

* liver decompensation child younger than 3 years patients with hepatitis B infection contraindications to perform MRI (intraocular metallic foreign body, cardiac pacemaker, intracranial clips of arterial brain aneurysms) refusal to participate in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
liver iron concentration using magnetic resonance imaging (T2* gradient echo pulse sequence in the axial plane) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt